CLINICAL TRIAL: NCT01521533
Title: A Multi-center, Open Label, Uncontrolled, Phase IIA Clinical Trial Evaluating the Safety and Efficacy of NOX A12 in Combination With a Background Therapy of Bortezomib and Dexamethasone (VD) in Previously Treated Patients With Multiple Myeloma (MM)
Brief Title: NOX-A12 in Combination With Bortezomib and Dexamethasone in Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNOXA12C301; 2011-004651-40 (EudraCT Number)
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Multiple Myeloma; NOX-A12; Velcade; Dexamethasone; Spiegelmer; Chemosensitization; Stromal cell-derived factor-1 (SDF-1); CXCL12
MeSH Terms: conditions — Multiple Myeloma | interventions — NOX-A12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NOX-A12 (Experimental)
  Interventions: Drug: NOX-A12

INTERVENTIONS:
Drug: NOX-A12 — Pilot Group (NOX A12 single agent, and combined with VD):
  * 3 cohorts of 3 patients will receive treatment with NOX A12 alone at a single dose of 1, 2 or 4 mg/kg i.v. 2 weeks before the combination treatment of NOX A12 and VD will start. The combination of NOX A12 and VD will follow a dose titration design beginning at 1 mg/kg NOX A12 (cycle 1) proceeding to dose levels of 2 mg/kg (cycle 2) and 4 mg/kg (cycle 3) NOX A12 in combination with VD. This is followed by consolidation in cycles 4-8 when NOX-A12 will be kept at the highest individually titrated dose.
  Expansion Group (NOX A12 in combination with VD):
  * Expansion patients will not receive single agent NOX-A12, but will receive combination treatment as for the pilot group.
  Other Names: olaptesed

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of NOX A12 alone and in combination with a background therapy of bortezomib and dexamethasone (VD) chemotherapy in previously treated patients with multiple myeloma (MM).

DETAILED DESCRIPTION:
Malignant plasma cells express high levels of CXCR4 chemokine receptors, which cause cell migration and adhesion to stromal cells secreting the CXCR4 ligand, CXCL12 (SDF-1). NOX A12 is a specific CXCL12 antagonist and may improve chemotherapy by disrupting CXCR4-CXCL12 interactions, thereby mobilizing plasma cells from protective tissue microenvironments to the blood. Furthermore, SDF-1 inhibition may alter the activation status of plasma cells, thereby triggering apoptosis or sensitization of plasma cells towards chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years.
2. Diagnosis of relapsed multiple myeloma for which bortezomib/dexamethasone would be given as standard of care.
3. Bortezomib-naïve or bortezomib-sensitive patient (i.e. best response of PR or better, sustained for at least 6 months), who did not receive bortezomib during the last line of therapy for MM prior to this study.
4. Progressive disease according to International Myeloma Working Group criteria.
5. Pre-study WHO Performance Status ≤ 2 and modified CIRS score of less than 7.
6. Signed and dated, written informed consent.
7. Men and women of reproductive potential must agree to follow accepted contraception methods during treatment and for 3 months after completion of treatment.
8. Acceptable liver function: Bilirubin ≤ 1.5 x upper limit of normal (ULN).
9. Acceptable hematology and hemostasis status: Platelet count ≥ 75 x 109/L, ANC > 0.75x109/L.
10. Acceptable renal function: Serum creatinine ≤1.5 ULN and/or calculated creatinine clearance ≥ 50 mL/min (calculated according to Cockroft & Gault formula).
11. No clinically significant abnormalities of liver volume, liver hemodynamics or elasticity, measured by abdominal ultrasound.

Exclusion Criteria:

1. The patient has a history of, or is clinically suspicious for, cancer-related Central Nervous System disease.
2. Prior allogeneic stem cell transplant (alloSCT) or patients who are considered to be candidates for alloSCT as assessed by their treating physician.
3. Patient has a history of other active malignancies within 3 years prior to study entry, with the exception of: adequately treated in situ carcinoma of the cervix uteri; basal or squamous cell carcinoma of the skin; in situ carcinoma of the bladder; previous malignancy confined and surgically resected with curative intent.
4. The patient exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to: uncontrolled systemic infection (viral, bacterial, or fungal); diagnosis of fever and neutropenia within 1 week prior to study drug administration.
5. Female patient is pregnant or breast-feeding.
6. Known infection with HIV, active Hepatitis B or Hepatitis C.
7. The patient has a history of prior toxicity from bortezomib or dexamethasone that resulted in permanent discontinuation of respective treatments.
8. Clinical evidence of a current significant (grade 2 or higher) or progressive neuropathy.
9. Treatment with any other investigational agent, or participation in another clinical trial within 30 days prior to study drug administration.
10. Uncontrolled hypertension (defined as systolic blood pressure [BP] > 160 mm Hg or diastolic BP > 100 mm Hg).
11. Myocardial infarction or unstable angina within the past 6 months prior to study drug administration. Heart failure of New York Heart Association functional Class III or IV prior to study drug administration.
12. Evidence of bleeding diathesis (greater than normal risk of bleeding) or coagulopathy (in the absence of therapeutic anticoagulation).
13. Systemic illnesses or other severe concurrent disease or alcoholism, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and efficacy of the investigational treatments.
14. Known or suspected of not being able to comply with the trial protocol.
15. Having been previously enrolled in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR = best response at least partial response (PR)) | 6 months
  Assessment of the overall tumor response after cycle 4 and 8 will be the primary efficacy endpoint. The recommendations for the uniform reporting of clinical trials as published by the International Myeloma Workshop Consensus Panel 1 in 2011 will be applied.
Safety and tolerability of NOX A12 alone and in combination with VD | 18 months
  The safety evaluation will be based on the following assessments:
  * Adverse events
  * Vital signs
  * 12 lead ECGs
  * Laboratory parameters
  * Abdominal ultrasound
  * Immunogenicity

SECONDARY OUTCOMES:
Effect of NOX A12 alone and combined with VD on the mobilization of peripheral blood CD34+ cells, plasma cells and myeloma cells | 6 months
Additional response criteria such as Minor Response (MR), immunophenotypic Complete Response and molecular Complete Response | 6 months
Time to event endpoints such as Progression Free Survival (PFS), Time To Progression (TTP) and Duration Of Response (DOR) following treatment with NOX A12 in combination with VD | 18 months
Plasma concentration of SDF-1 after treatment with NOX-A12 alone (pilot group only) and in combination with VD | 6 months
Pharmacokinetics of NOX A12 alone (pilot group only) and combined with VD | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kai Riecke, MD, Study Director — TME Pharma AG
Locations (10):
- Austria (2):
  - University Hospital Salzburg, Department of Medicine III, Center of Oncology and Hematology, Salzburg
  - Wilhelminenspital, Department of Medicine I, Center of Oncology and Hematology, Vienna
- France (2):
  - Hôpital Huriez, Centre Hospitalier Régional Universitaire de Lille, Lille
  - Hôpital Saint Antoine - Service des maladies du sang et de thérapie cellulaire, Paris
- Germany (3):
  - University Hospital Freiburg, Medizinische Universitätsklinik, Innere Medizin I, Haematologie und Onkologie, Freiburg im Breisgau
  - University Hospital Münster, Medizinische Klinik und Poliklinik A, Münster
  - University Hospital Ulm, Zentrum für Innere Medizin,, Ulm
- Italy (3):
  - University Hospital San Martino, Department of Hematology and Oncology, Genova
  - Niguarda Ca'Granda Hospital, Department of Hematology, Milan
  - Sapienza University of Rome, Department of Hematology, Rome

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581